CLINICAL TRIAL: NCT07301866
Title: Single-site, Prospective, Open-label Phase I-II Study on Transplantation Using Cord Blood Treated With an Optimized Dose of UM171: Optimized ECT-001-CB.
Brief Title: A Study Testing an Improved Dose of UM171 to Help Make Cord Blood Transplants More Effective and Safe.
Acronym: ECT-001-CB-013
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ciusss de L'Est de l'Île de Montréal (Other)
Collaborators: Stem Cell Network (Other)
Responsible Party: Principal Investigator, Sandra Cohen, Dr., Ciusss de L'Est de l'Île de Montréal
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ECT-001-CB-013
Record Dates: First submitted 2025-11-27; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Acute Leukemia, High Risk; Myelodysplastic Syndromes, High Risk; Hematologic Malignancy Requiring an Allogeneic Hematopoietic Stem Cell Transplant Lacking a Donor
Keywords: High risk hematologic malignancy; Cord blood transplant; UM171; ECT-001-CB; Lack of donor for stem cell transplant donor; Acute leukemia; Myelodysplastic syndrome
MeSH Terms: conditions — Myelodysplastic Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- UM171 CB transplant (ECT-001-CB) with optimized dose of UM171 (Experimental)
  Interventions: Biological: ECT-001-CB

INTERVENTIONS:
Biological: ECT-001-CB — UM171-expanded cord blood

SUMMARY:
This clinical study is testing a new way to improve stem cell transplants for adults with high-risk blood cancers, such as leukemia or myelodysplasia, who do not have a suitable donor. The transplant uses stem cells from umbilical cord blood that have been expanded in the lab using a molecule called UM171. Previous studies showed that UM171 helps these cells grow and work better, leading to faster blood count recovery and fewer complications.

In this study, researchers are testing whether increasing the dose of UM171 during the lab expansion process can make the transplant less toxic. The hypothesis is that using a higher dose of UM171 to expand cord blood stem cells will help patients recover blood counts faster after transplant by improving the growth and function of the cells. This may lead to better immune recovery, fewer infections, shorter hospital stays, and improved overall outcomes.

Only seven patients will be enrolled, and they will be followed for one year after their transplant.

DETAILED DESCRIPTION:
This is a single-center, prospective, open-label, dose-escalating Phase I/II clinical trial designed to evaluate the safety, feasibility, and efficacy of ECT-001-CB cord blood transplantation using an optimized dose of UM171, a small molecule that enhances hematopoietic stem cell (HSC) expansion.

Allogeneic hematopoietic stem cell transplantation (HSCT) is a potentially curative treatment for patients with high-risk hematologic malignancies. However, some patients lack a suitable donor. Cord blood (CB) is a valuable alternative donor source due to its tolerance for HLA mismatches and lower incidence of chronic graft-versus-host disease (GVHD). Despite these advantages, CB transplantation has declined due to limitations such as low cell dose, delayed engraftment, and increased non-relapse mortality (NRM).

UM171 is a proprietary molecule that has demonstrated the ability to expand CD34⁺ HSCs ex vivo, thereby addressing the cell dose limitation of CB transplants. Previous trials using UM171-expanded CB units (ECT-001-CB) showed promising results, including faster engraftment, improved immune reconstitution, and reduced NRM.

This study builds on prior findings by investigating whether a higher dose of UM171 (125nM vs. the conventional 35nM) can further accelerate neutrophil engraftment and enhance immune recovery. Preclinical data suggest that higher UM171 concentrations may increase the number of long-term repopulating HSCs and promote balanced lymphoid and myeloid differentiation, potentially improving clinical outcomes.

Seven patients with high-risk acute leukemia or myelodysplasia, or other hematologic malignancies requiring HSCT and lacking a suitable donor, will be enrolled over a 12-month period. Patients will receive a single ECT-001-CB transplant following an intermediate or high-intensity conditioning regimen. The CB unit will be expanded ex vivo with escalating doses of UM171 (starting at 70nM, potentially increasing to 125nM based on engraftment outcomes).

Primary endpoints include safety (grade ≥3 adverse events), feasibility of manufacturing and infusion, and time to neutrophil engraftment. Secondary endpoints include NRM, platelet engraftment, graft failure, progression-free survival (PFS), overall survival (OS), incidence of acute and chronic GVHD, immune reconstitution, and time to hospital discharge. Exploratory endpoints include infectious complications, relapse incidence, GVHD-free relapse-free survival (GRFS), advanced immunologic profiling, and comparisons with historical controls.

Safety will be monitored by an independent Data Safety Monitoring Board (DSMB). The study includes predefined stopping rules to ensure patient safety, including thresholds for engraftment delay, graft failure, NRM, and severe GVHD.

This trial aims to optimize CB transplantation by enhancing the efficacy of UM171-expanded grafts, potentially offering a safer and more effective treatment option for patients with limited donor availability.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects ≥ 18 and ≤ 67 years old,
2. Patient with either i. High risk acute leukemia or myelodysplasia defined as expected 2 year OS or PFS < 40% after a conventional allogeneic HSC transplant or ii. A hematologic malignancy requiring an allogeneic hematopoietic stem cell transplant and lack of a suitable HLA identical, haploidentical or 7/8 HLA matched donor.
3. Availability of an adequate CB for expansion:

   i. ≥ 5/8 HLA match when A, B, C and DRB1 are performed at the allele level.

   ii. Minimal cell dose: TNC ≥ 1.5 x 107/kg, and CD34 ≥ 0.5 x 105/kg. iii. Needs to be erythrodepleted by bank prior to cryopreservation. iv. Must comply with local site regulations AND, come from a cord bank that is FACT, or AABB accredited, or FDA approved or eligible for NMDP IND (unless PI approves another bank).

   v. To meet eligibility criteria, the patient's weight at time of cord selection will be used; however, if this weight has increased by more than 5% at time of admission to hospital and with the new weight the patient no longer meets eligibility criteria for cell dose, LI approval will be required to move forward with the selected cord. Every attempt will be made to always use the most recent weight in cord selection
4. Patients with adequate physical function as measured by:

   i. Karnofsky score ≥ 70% ii. Hematopoietic comorbidity index (HCT-CI): 0-3 for 2nd transplant and age 60-65 years, 0-5 if <60 years old, and 0-2 if 66-67 years.

   iii. Adequate cardiac function: Left ventricular ejection fraction ≥ 40% within 60 days prior to start of conditioning regimen iv. Adequate pulmonary function: Forced vital capacity (FVC), forced expiratory volume in 1 second (FEV1) and diffusing capacity corrected for hemoglobin (DLCOc) ≥ 50% of predicted within 60 days prior to start of conditioning regimen.

   v. Adequate hepatic function: Bilirubin < 2 x ULN unless felt to be related to Gilbert's disease or hemolysis; AST and ALT ≤ 2.5 x ULN (the PI may approve up to 3 times ULN) ; alkaline phosphatase ≤ 5 x ULN.

   vi. Adequate renal function: Estimated or measured creatinine clearance ≥ 60 ml/min/1.73m2.
5. A back up graft must have been identified prior to initiation of conditioning regimen.
6. Signed written informed consent.
7. Female patients of childbearing potential must have a negative serum pregnancy test within 30 days of enrolment and within 30 days of starting of preparative regimen; patient must be willing to use an effective contraceptive method while enrolled in the study.

Exclusion Criteria:

1. Allogeneic or autologous myeloablative transplant within last 6 months.
2. Patients with inadequate physical function as measured by:

   i. Active, uncontrolled bacterial, viral or fungal infection (currently taking medication with evidence of either progression of clinical symptoms or radiologic findings or lack of evidence of response to therapy).

   ii. Presence of a malignancy other than the one for which the HSC transplant is being performed, with an expected survival estimated to be less than 75% at 5 years.

   iii. Seropositivity for HIV. iv. Hepatitis B or C infection with measurable viral load. Patients with hepatitis B or C infection regardless of viral load require clear documentation of absence of cirrhosis by either fibroscan or biopsy.

   v. Liver cirrhosis.
3. Positive anti-donor HLA antibodies with MFI above 1500 against the selected CB (PI may approve an MFI up to 5000; if above 2500, desensitization is strongly recommended)
4. Use of an investigational agent within 30 days (defined as a drug not approved by Health Canada or FDA regardless of indication) of start of chemotherapy unless documented approval obtained from Sponsor.
5. Presence of ≥30% blasts in bone marrow or ≥ 0.5 x109/L blasts in circulating blood
6. Active central nervous system involvement or chloroma > 2 cm.

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Estimated)
Dates: Start 2025-10-06 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Incidence of grade 3 or higher adverse events (AEs) | From the start of pre-transplant conditioning of first patient throught 1 year post-transplant of last patient
  Incidence of grade 3 or higher adverse events (AEs)
Feasibility of manufacturing and infusion | From first day of product manufacturing for the first patient throught the infusion of the product to the last patient, up to Month 13.
  Proportion of selected grafts that will be expanded and meet release criteria and be successfully infused to the patient
Time to neutrophil engraftment | From day of transplant (Day 0) throught day of neutrophil engraftment, up to Day 42 post-transplant.
  Neutrophil engraftment is defined as the first day of neutrophil count (ANC) ≥ 0.5 x 109/L for 3 consecutive days; first day of ANC ≥ 0.1 x 109/L will also be documented.

SECONDARY OUTCOMES:
Incidence of NRM at 1 year post transplant | From day of transplant (Day 0) of first patient throught 1 year post-transplant of last patient
  Defined as death not preceded by recurrent or progressive malignancy occurring anytime after stem cell infusion
Time to platelet engraftment | From day of transplant (Day 0) throught day of platelet engraftment, up to Day 42 post-transplant.
  Platelet engraftment is defined as the first of 3 days of a sustained platelet count ≥ 20 x 109/L with no platelet transfusion in the preceding 7 days as per CIBMTR standards.
Incidence of graft failure | From day of transplant (Day 0) of first patient throught 1 year post-transplant of last patient
  The incidence of graft failure will be monitored throughout the protocol until 1 year post transplant
Progression-free survival (PFS) at 1 year post-transplant | From day of transplant (Day 0) of first patient throught 1 year post-transplant of last patient
  Relapse/progression is defined by either hematologic or extramedullary evidence of disease.
Overall Survival (OS) at 1 year post-transplant | From day of transplant (Day 0) of first patient throught 1 year post-transplant of last patient
  OS is defined as the time interval between day of transplant until death from any cause or for surviving patients, to last follow-up. An event is defined as death from any cause
Incidences of grade 2-4, 3-4 acute and moderate-severe chronic GVHD at 1 year | From day of transplant (Day 0) of first patient throught 1 year post-transplant of last patient
  Standard clinical criteria and histologic evaluation when possible of skin, liver or gastrointestinal tract will be used to establish and grade acute GVHD. The time to onset of acute GVHD grade 2-4 and maximal grade will be recorded. More specifically, time of onset to grade 2 GVHD as well as time of onset of grade 3 or 4 acute GVHD will be collected.
  Cumulative incidence of moderate-severe chronic GVHD will be determined at 12 months. Chronic GVHD will be diagnosed and graded according to the recommendations of the NIH Consensus Conference and recently updated.
Immune reconstitution at 2, 3, 6 and 12 months | From day of transplant (Day 0) of first patient throught 1 year post-transplant of last patient
  CD4+, NK and B cell counts (T-B-NK panel) and IgG levels will be measured at 2, 3, 6, and 12 months post-transplant. These results may be compared to conventional dose ECT-001-CB transplants or other types of transplant.
Time to discharge from hospital | From day of transplant (Day 0) of first patient throught 1 year post-transplant of last patient
  Duration of initial transplant hospitalization will be measured from day of transplant until day of hospital discharge. These results may be compared to various control groups

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Cohen, Dr., Principal Investigator — CIUSSS de l'Est-de-l'Ile-de-Montréal
Locations (1):
- Hôpital Maisonneuve-Rosemont, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
Description:
  The sponsor plans to share IPD collected during the trial, including de-identified clinical data and biological sample results, with qualified researchers for secondary analyses. This includes data related to:
  Primary and secondary endpoints (e.g., neutrophil engraftment, GVHD incidence, survival outcomes) Safety data (e.g., adverse events, serious adverse events) Demographic and baseline characteristics
  What IPD Will Be Shared:
  * De-identified individual-level clinical data
  * Immune profiling and chimerism data
  * Adverse event and safety data
  * Outcome measures (e.g., engraftment times, relapse, survival)
Supporting Information: Study Protocol, CSR
Time Frame: IPD will be available after the completion of the study and publication of primary results, estimated to be within 12 months following the final patient's last follow-up visi
Access Criteria: A proposal that describes planned analyses must be submitted to the Principal Investigator, Dr. Sandra Cohen, and a data sharing agreement must be signed.